CLINICAL TRIAL: NCT02694406
Title: Added Value of MRI Perfusion in Evaluation of Complex Adnexal Masses
Brief Title: MRI Perfusion in Adnexal Masses
Acronym: MRI-CAM
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: MRI-CAM
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Complex Adnexal Masses
Keywords: Diagnosis
MeSH Terms: conditions — Disease | interventions — Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: MRI perfusion — contrast-enhanced MR imaging including perfusion weighted imaging (PWI)

SUMMARY:
As ovarian cancer is characterized by an anarchic neovascularization resulting in a wide number of immature microvessels. These vessels are characterized by a lack of coverage by pericytes and the higher expression of one of the receptors of Vascular Endothelial Growth Factor on both endothelial and epithelial cells of ovarian cystadenocarcinomas. These physio pathogenic characteristics have been demonstrated to be in line with variations of MR perfusion parameters.

Unlike many lesions that occur in other parts of the body, biopsy should not be performed in adnexal masses that demonstrate no evidence of peritoneal disease because it may cause spillage of cystic contents, potentially leading to iatrogenic up-staging of what may have been a malignant tumor that was limited.

ELIGIBILITY:
Inclusion Criteria:

* complex adnexal mass
* patient fit for surgery

Exclusion Criteria:

* any general contraindication to MRI
* severely ill patients
* those with claustrophobia.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with adenxal masses
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
detect the number of malignant adnexal masses | 2 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ahmed Abbas, Assiut, Cairo Governorate
  - Ahmed Abbas, Asyut

IPD SHARING:
Plan to Share IPD: Undecided